CLINICAL TRIAL: NCT01393288
Title: Developing Individualized Strategies to Prevent Nausea and Vomiting
Acronym: PDNVF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1R01CA163074-01A1; 10831533 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Postoperative Nausea and Vomiting; Genetic Polymorphisms
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron; Lorazepam; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ondansetron (Placebo Comparator)
  Interventions: Drug: Ondansetron
- Lorazepam (Placebo Comparator)
  Interventions: Drug: Lorazepam
- Aprepitant (Placebo Comparator)
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Ondansetron — 8 mg ondansetron ODT or placebo, 1 hour pre-operatively, before discharge, evening of day of surgery, morning of postoperative day (POD) 1, lunch POD 1, evening POD 1, and morning of POD 2
  Arms: Ondansetron
Drug: Lorazepam — 1 mg Lorazepam or placebo 1 hour preoperatively, before discharge, evening of day of surgery, morning of postoperative day (POD) 1, lunch of POD 1, evening of POD 1, and morning of POD 2.
  Arms: Lorazepam
Drug: Aprepitant — 40 mg Aprepitant or placebo 1 hour preoperatively and before discharge (placebo for postoperative days 1-2)
  Arms: Aprepitant

SUMMARY:
Every year, more than 5 million patients in the US experience postoperative nausea and/or vomiting (PONV) and in the ambulatory setting post-discharge nausea and/or vomiting (PDNV) is the most common cause for unanticipated hospital re-admissions. Similarly, millions of patients suffer from chemotherapy induced nausea and/or vomiting (CINV), and one out of five patients discontinues chemotherapy for this reason. Thus, the control of nausea and vomiting remains a major health concern for the investigators society. The investigatorsoverall goal is to further the understanding of nausea and vomiting and optimize antiemetic selection in order to facilitate individualized patient care.

Unfortunately, current antiemetics reduce the incidence of nausea by only about one third. As a result, antiemetics are often combined, exposing patients to adverse events and drug interactions without evidence for the most effective combination. Moreover, it remains unclear why such a large amount of inter-individual variability exists in antiemetic responsiveness. 5HT3, NK1, and GABA receptors are targets for some of the most commonly prescribed anti-emetics. Furthermore, these receptors have many known genetic polymorphisms, including several linked to incidence of nausea and vomiting. Thus pharmacogenomic variation may in part explain interindividual differences in treatment responses and will be tested in this proposal.

Leveraging the established infrastructure of the UCSF Clinical and Translational Science Institute, and the support of 6 patient recruitment sites, the investigators will enroll 1280 high risk patients to three oral interventions with distinct mechanisms of action for nausea and vomiting. Investigating nausea and vomiting in ambulatory surgical patients is an excellent model for this trial owing to a high incidence, short observational period, and the ability to standardize and control potentially confounding variables. In this proposal, 100% of patients will receive a single intraoperative dose of 4 mg ondansetron, which is similar to the 80% of patients who receive prophylaxis in common practice. Using a factorial design, these patients will be randomized to receive one out of eight possible combinations of the three interventions (ondansetron, aprepitant, lorazepam) versus placebo (ond+aprep+lora, ond+aprep, ond+lora, aprep+lora, ond, aprep, lora, or placebo). Thus, in this proposal 87.5% (7 out of 8 patients) will have antiemetic coverage for the postdischarge period, which is considerably higher than in common practice, where only 4% of patients have antiemetic coverage after discharge. The primary endpoint will be the prevention of nausea and vomiting within 48 hours after ambulatory surgery. The advantage of the factorial trial design is its high efficiency to systematically investigate multiple interventions while allowing us to test for potential interactions. It is also an ideal format for the simultaneous assessment of pharmacogenomic interactions of antiemetics in this proposal.

To this end, the investigators will collect DNA samples and take advantage of the unique opportunity to investigate the effects of variation in candidate receptor genes in the context of the three treatment interventions for PDNV. This approach may in part explain inter-individual differences in drug efficacy and allow for future screening of at-risk patients. Specifically, the investigators will be assessing single nucleotide polymorphisms (SNPs) and copy number variants (CNVs) of targeted receptors for the antiemetics tested.

Aim 1: To determine efficacy of three interventions for the prevention of PDNV.

Hypothesis 1.1: Each intervention reduces the incidence of PDNV.

Hypothesis 1.2: Efficacy of all interventions is independent so that efficacy of a combination can be derived from the efficacy of the individual interventions.

Aim 2: To determine if drug response for anti-emetics is dependent upon genetic variance.

Hypothesis 2: Efficacy of ondansetron, aprepitant and lorazepam to reduce PDNV differs with 5HT3, NK1, and GABA receptor gene variation, respectively.

ELIGIBILITY:
Inclusion Criteria:

* adult (i.e. at least 21 years of age) ambulatory surgery patients, with a duration of 1-4 hours
* able to understand, read, and write in English, are ASA physical status 1-3, and are high risk PDNV patients (with 3 or more of the following risk factors:
* female gender
* age < 50
* history of PONV and/or currently prone to motion sickness, and expectation of post-op opioid use).

Exclusion Criteria:

* patients not at high risk for PDNV (as described above)
* patients <21 years of age
* planned inpatient surgical patients
* planned total intravenous anesthesia, sedation, or regional technique without inhaled anesthetic
* inability to provide informed consent in English
* pregnant or breastfeeding
* persistent and/or current nausea/vomiting.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11; Study Completion 2015-11

PRIMARY OUTCOMES:
Incidence of post-discharge nausea and vomiting (PDNV) | 48 hours post-discharge

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Hospital, Lexington, Kentucky
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio